CLINICAL TRIAL: NCT04681586
Title: Bright Light Therapy as Possible Treatment Option for Fatigue in Multiple Sclerosis Patients - A Randomised Controlled Trial
Brief Title: Bright Light Therapy as Possible Treatment Option for MS-Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: National Bank of Austria (Other Government)
Responsible Party: Principal Investigator, Stefan Seidel, Associate Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP18005ONB
Record Dates: First submitted 2020-10-20; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: bright light therapy; MS-Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright white light (Experimental)
  Interventions: Device: bright light therapy
- Dim red light (Placebo Comparator)
  Interventions: Device: dim red light

INTERVENTIONS:
Device: bright light therapy — using a bright light therapy device (10.000 lux) for 30min every morning for two weeks
  Arms: Bright white light
Device: dim red light — using the same device as the active group, but with an installed filter that dims light to <300 lux for 30min every morning for two weeks
  Arms: Dim red light

SUMMARY:
This study aims to investigate the effect of a 2-week trial of bright light therapy (BLT, 10.000 lx) on fatigue in multiple sclerosis (MS) patients. In this randomised placebo-controlled trial, the effect of bright light therapy will be compared to dim red light. MS-fatigue is quantified by patients using a visual analogue scale (VAS) and activity levels, subjective and objective sleep parameters and daytime sleepiness are measured.

DETAILED DESCRIPTION:
Materials and methods:

* visual analogue scale (4x/day for 6 weeks; measuring fatigue)
* wrist actigraphy (6 weeks)
* sleep diaries (6 weeks)
* polysomnography (2x)
* multiple sleep latency test (2x)
* 4 subtests of the TAP (Testbatterie zur Aufmerksamkeitsprüfung; Alertness, Vigilance, Go/No-Go, Split Attention)
* questionnaires (Fatigue Severity Scale, Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index, Beck Depression Inventory, Beck Anxiety Inventory, Modified Fatigue Impact Scale, Morningness-Eveningness Questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* MS patients who suffer from fatigue
* Age between 18 and 65 years old
* FSS Score of 36 or greater
* ESS Score of 12 or greater
* MEQ Score between 31 and 69
* BDI Score lower than 19
* BAI Score lower than 27
* EDSS lower than 4

Exclusion Criteria:

* sleep disorders (periodic limb movement disorders, obstructive or central sleep apnea, REM sleep behavior disorders)
* change of antidepressive/fatigue influencing/sleep influencing/photosensizing/MS medication within the preceding 4 weeks
* clinical MS-relapse within the preceding 4 weeks
* consumption of alcohol: more than 1 glass per day
* consumption of caffeine: more than 4 cups per day
* current shift work
* Jet lag (travelled across two or more time zones within 90 days before study screening
* Retinopathy or other visual diseases/abnormalties
* Traumatic brain injury within the preceding 5 years
* pregnant or lactating
* Participation in another clinical trial at the same time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue levels | Day 1, Day 14, Day 30, Day 46
  Improvement of MS-fatigue symptoms as measured with questionnaires (Fatigue Severity Scale; FSS, Modified Fatigue Impact Scale; MFIS and a visual analogue scale)
Change in fatigue levels | Day 15, Day 31
  Improvement of MS-fatigue symptoms as measured with psychological testing (Testbatterie zur Aufmerksamkeitsprüfung; TAP)

OTHER OUTCOMES:
Change in nighttime sleep | Day 14, Day 30
  Improvement in nighttime sleep as measured with polysomnography (PSG)
Change in daytime sleepiness | Day 15, Day 31
  Improvement of sxcessive daytime sleepiness as measured using a multiple sleep latency test (MSLT) and Epworth Sleepiness Scale (ESS)
Change in activity levels | Day 1 through day 46
  Rapprochement of activity levels according to circadian rhythms
Change in psychological well-being | Day 1, Day 14, Day 30, Day 46
  Improvement in depression and anxiety scores as measured by Beck Depression Inventory (BDI) and Beck Anxiety Inventory (BAI)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided